CLINICAL TRIAL: NCT03040986
Title: A Phase II Study of Selumetinib (AZD6244) for the Treatment of Advanced Pancreas Cancer Harboring KRAS G12R Mutations
Brief Title: Selumetinib Sulfate in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer With KRAS G12R Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00118; NCI-2017-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17C0144; 10050 (Other: National Cancer Institute LAO); 10050 (Other: CTEP); ZIABC011078 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: KRAS NP_004976.2:p.G12R; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IV Pancreatic Cancer AJCC v6 and v7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selumetinib sulfate) (Experimental): Patients receive selumetinib sulfate by mouth (PO) twice daily (BID). Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib Sulfate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib Sulfate — Given by mouth (PO)
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Selumetinib Sulphate

SUMMARY:
This phase II trial studies how well selumetinib sulfate works in treating patients with pancreatic cancer with Kirsten rat sarcoma (KRAS) G12R mutations that has spread from where it started to nearby tissue or lymph nodes or other places in the body. Selumetinib sulfate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate to selumetinib sulfate (selumetinib) administered as 75 mg orally twice daily on a continuous schedule in patients with advanced pancreas cancer harboring Kirsten rat sarcoma (KRAS) G12R mutations.

SECONDARY OBJECTIVES:

I. To determine the progression free survival of patients with locally advanced, unresectable and stage IV pancreas cancer treated with selumetinib monotherapy.

II. To evaluate the safety of selumetinib in patients with advanced pancreas cancer.

III. To determine the impact of additional genetic alterations on the response to selumetinib in pancreas cancer harboring KRAS G12R mutations.

IV. To develop a clinically applicable biomarker predicting response to selumetinib in pancreas cancer harboring KRAS G12R mutations.

OUTLINE:

Patients receive selumetinib sulfate orally (PO) twice daily (BID). Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed locally advanced or metastatic pancreas cancer
* Patients must have received at least 6 months fluorouracil (5-FU)- or gemcitabine-based treatments for pancreas cancer (fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin [FOLFIRINOX], fluorouracil, leucovorin calcium and oxaliplatin [FOLFOX], 5-FU+ nal-IRI [MM-398; nanoliposomal irinotecan], or 5-FU [including capecitabine], gemcitabine-based gemcitabine plus abraxane, gemcitabine monotherapy among others)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have Clinical Laboratory Improvement Act (CLIA) confirmed somatic Kirsten rat sarcoma (KRAS) G12R mutation as determined by sequence analysis of matched normal deoxyribonucleic acid (DNA) from any specimen obtained from the individual; patients must provide tumor sample for KRAS analysis or be willing to undergo mandatory screening biopsy
* Patients must not have had chemotherapy, molecular therapy with erlotinib, radiation therapy, or experimental biological or molecular therapy for at least 4 weeks prior to starting study medication; patients who received FOLFIRINOX must be 6 weeks from the last administration of therapy; patients must have recovered from any acute toxicity related to prior therapy or surgery, to a grade 1 or less unless specified
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 or Karnofsky >= 70%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin (Hgb) >= 9.0 g/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 3 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR
* Creatinine clearance > 60 mL/min/1.73 m^2 by either Cockcroft-Gault formula or 24-hour urine collection analysis
* Patients must be willing to return to the clinic for follow-up visits
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 weeks after dosing with selumetinib sulfate (AZD6244) ceases; women of child-bearing potential must have a negative pregnancy test within 14 days prior to study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform her treating physician immediately; please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 12 weeks post-last dose due to sperm life cycle; NOTE: breastfeeding should be discontinued if the mother is treated with selumetinib
* Ability to understand and the willingness to sign a written informed consent document or patients with Impaired Decision Making Capacity (IDMC) if they are represented by a Legally Authorized Representative (LAR)
* Patient must be able to reliably swallow oral medications

Exclusion Criteria:

* Patients who have received prior treatment with tyrosine kinase inhibitors (e.g. erlotinib), or anti-Epidermal growth factor receptor (EGFR) agents (e.g. cetuximab, panitumumab)
* Patients currently receiving any medication known to induce central serous chorioretinopathy which in the opinion of the principal investigator, would make the administration of study drug hazardous
* Patients with active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any underlying medical condition which, in the opinion of the principal investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial; no additional workup is needed to exclude brain metastases if the patient is asymptomatic or has no history of brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Selumetinib (AZD6244) or other agents used in study
* Previous Mitogen-activated protein kinase kinase (MEK), RAS, or Rapidly Accelerated Fibrosarcoma (RAF) inhibitor use
* Patients with the following cardiac conditions are excluded:

  * Uncontrolled hypertension (blood pressure [BP] of >= 150/95 despite medical support/management)
  * Acute coronary syndrome within 6 months prior to starting treatment
  * Uncontrolled angina - Canadian Cardiovascular Society grade II-IV despite medical support/management
  * Heart failure New York Heart Association (NYHA) class II or above
  * Prior or current cardiomyopathy (within 6 months) including but not limited to the following:

    * Known hypertrophic cardiomyopathy
    * Known arrhythmogenic right ventricular cardiomyopathy
    * Abnormal ejection fraction (echocardiogram [ECHO]) =< 53% (if a range is given then the upper value of the range will be used) or cardiac magnetic resonance imaging (MRI)
    * Previous moderate or severe impairment of left ventricular systolic function (left ventricular ejection fraction [LVEF] < 45% on echocardiography or equivalent on multi-gated acquisition scan [MUGA]) even if full recovery has occurred; echocardiogram (Echo) and additional cardiac studies not indicated unless clinically symptomatic or patient has significant cardiac history
    * Severe valvular heart disease
    * Atrial fibrillation with a ventricular rate > 100 beats per minute (bpm) on electrocardiogram (ECG) at rest
    * Fridericia's corrected QT interval (QTcF) >= 450 msec or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) are excluded; the use of medication(s) that can prolong QTc interval is prohibited while treated on this study
* Patients with known ophthalmologic conditions, such as:

  * Current or past history of central serous retinopathy
  * Current or past history of retinal vein occlusion
  * Known intraocular pressure (IOP) > 21 mmHg (or upper limit of normal [ULN] adjusted by age) or uncontrolled glaucoma (irrespective of IOP); patients with controlled glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) may be eligible after discussion with the study chair
  * Subjects with any other significant abnormality on ophthalmic examination (performed by an ophthalmologist) should be discussed with the study chair for potential eligibility
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal plexiform neurofibroma (PN) (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Patients with refractory nausea and vomiting, chronic gastrointestinal (GI) diseases (e.g., inflammatory bowel disease) or significant bowel resection
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; HIV-positive patients not on antiviral therapy with undetectable viral loads and cluster of differentiation 4 (CD4) counts > 300, and after confirmation of eligibility after discussing with the study chair are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, Principal Investigator — National Cancer Institute LAO
Locations (9):
- United States (9):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenney C, Kunst T, Webb S, Christina D Jr, Arrowood C, Steinberg SM, Mettu NB, Kim EJ, Rudloff U. Phase II study of selumetinib, an orally active inhibitor of MEK1 and MEK2 kinases, in KRASG12R-mutant pancreatic ductal adenocarcinoma. Invest New Drugs. 2021 Jun;39(3):821-828. doi: 10.1007/s10637-020-01044-8. Epub 2021 Jan 6. PMID 33405090

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 180 pts were not enrolled to the study. All pts who made contact to participate in the study all had KRAS G12R mutation testing thus pre-screening was not necessary. The 1st 8 pts who made contact with the study and were eligible were consented, enrolled and treated. No other pts were enrolled in the study per the statistical design in the protocol. As pre-specified, the study did not move into the second phase due to lack of efficacy.
Groups:
- Dose Level 0: 75mg Selumetinib Sulfate Twice Daily: Participants receive 75mg selumetinib sulfate by mouth (PO) twice daily (BID). Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity.
- 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily: Participants receive 75mg selumetinib sulfate by mouth (PO) twice daily (BID) followed by 50mg twice daily. Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Started | 6 | 2
Completed | 0 | 0
Not Completed | 6 | 2
Not completed — Hospice | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Disease progression on study | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.99) | 59 (7.07) | 60.5 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8
Location of Primary Tumor [Count of Participants; unit: Participants]
  Head/Body | 4 | 1 | 5
  Tail | 2 | 1 | 3
Previous Treatments [Count of Participants; unit: Participants]
  Radiation | 2 | 1 | 3
  Surgery | 3 | 2 | 5
  Multiple agents systemic chemotherapy | 6 | 2 | 8
Number of Previous Lines of Systemic Chemotherapy [Number; unit: participants]
  1 | 1 | 0 | 1
  2 | 2 | 1 | 3
  ≥3 | 3 | 1 | 4
Number of Metastatic Sites (involved organs) [Number; unit: participants]
  1 | 2 | 0 | 2
  2 | 1 | 2 | 3
  ≥3 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an Objective Response (Partial Response + Complete Response)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm (<1 cm). Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately 1-8.2 months
Measure: Number; unit: Proportion of participants
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Proportion of participants
  Partial Response | 0 | 0
  Complete Response | 0 | 0

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first and was calculated using the Kaplan-Meier method.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 52 weeks
Population: All participants are grouped together as pre-specified in the protocol for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants: All participants that received 75mg selumetinib sulfate by mouth (PO) twice daily (BID); and 75mg Selumetinib sulfate twice daily followed by 50mg twice daily.
Arm/Group | All Participants
Number analyzed (Participants) | 8
Months | 3.0 [0.8 to 8.2]

3. Secondary Outcome: Incidence of Grade 3 or Greater Adverse Events Using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Probably or Definitely Attributable to the Agent Selumetinib
Description: Here are the grade 3 or greater adverse events assessed by the CTCAEv5.0 probably or definitely attributable to the agent Selumetinib. Grade 3 is defined as severe or medically significant, Grade 4 is life-threatening consequences, and Grade 5 is death related to adverse event. Probably is defined as likely related to the agent, and Definitely is defined as clearly related to the agent.
Time Frame: Date treatment consent signed to date off study, approximately 25 months and 6 days.
Measure: Number; unit: Adverse events
Groups:
- Probably Attributable: 75mg Selumetinib Sulfate Twice Daily: Participants receive 75mg selumetinib sulfate by mouth (PO) twice daily (BID). Treatment repeats every 28 days for up to 27 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Probably Attributable: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Adverse events
  Probably: Grade 3 Hypertension | 2 | 0
  Probably: Grade 3 Pancreatitis | 1 | 0
  Definitely: Grade 3 Alanine aminotransferase increased | 0 | 2
  Definitely: Grade 3 Dyspnea | 1 | 0
  Definitely: Grade 3 Heart failure | 1 | 0
  Definitely: Grade 3 Hypertension | 0 | 1

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 25 months and 6 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

5. Secondary Outcome: Semi-quantitative Measurements of Connector Enhancer of the Kinase Suppressor of Ras-1 (CNKSR1)
Description: Comparisons will be done to estimate the differences of the expression level in pancreas cancer tissues and clinical outcome variables.
Time Frame: Up to 52 weeks
Population: This outcome measure was not done because only 1 out of the 8 enrolled participants agreed to undergo biopsy while on treatment. Tumoral biopsies were not mandatory but optional for participants enrolled onto the study. Because only one biopsy specimen was obtained, on the discretion of the PI, no analysis and no comparisons were performed.
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Predictive Biomarkers for Response to Selumetinib
Description: Presence of variants identified in the 50-cancer gene panel will be compared with response, presenting the results in a 2x2 table with findings reported descriptively. Pre-treatment ctDNA levels will be divided into groups to separate aberrant values from the rest. The cutoffs will be > and < 2 standard deviations of the mean, with the cutoffs applied to both ctDNA levels. Based on these groups, resulting in participants with cell free deoxyribonucleic acid (cfDNA) transcripts levels > 2 standard deviation (SD) above the mean, participants with cfDNA transcripts levels < 2 SD below the mean, and the rest in between, the categorical results will be evaluated and reported relative to response vs. non-response in a descriptive manner.
Time Frame: Up to 52 weeks
Population: Since no responses were observed in either Arm/Group, the planned correlation was not conducted for this outcome measure.
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Longitudinal Biomarker Measuring Response to Treatment
Description: Circulating free deoxyribonucleic acid (cfDNA) transcript levels will be followed from the start of treatment every (q)2 weeks and the change to pre-treatment will be plotted for each timepoint in a spider plot format. Variant profile derived from voluntary repeat biopsies will be compared to pre-treatment variant profile and gain of variants (adjusted for similar sequencing depth) will be recorded.
Time Frame: start of treatment every (q)2 weeks, up to 52 weeks
Population: This outcome measure was not done because of the lack of ctDNA copy number determinations in participants on-treatment compared to pre-treatment levels in the participants whose ctDNA levels were longitudinally evaluable. No variant profiling of baseline tumoral tissues was performed.
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in the Somatic Circulating Tumor Deoxyribonucleic Acid (ctDNA) Mutation Profile and Its Correlation With Clinical Outcome
Description: The presence of mutant DNA copies and the fractional abundance of the mutant KRAS allele on circulating tumor DNA (ctDNA) in cell-free (cf) DNA isolated from plasma samples were to be determined.
Time Frame: Baseline up to 52 weeks
Population: No other somatic variants in ctDNA other than the KRAS allele were analyzed because the only available droplet digital PCR (ddPCR) assay was the one for the KRAS allele. Thus, the planned analysis change in the somatic ctDNA mutation profile and its correlation with clinical outcome was not conducted.
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Copy Number KRAS Wild Type Allele in Circulating Tumor DNA (ctDNA)
Description: ctDNA copy number measurements of KRAS wild type alleles in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples was determined from baseline and the last KRAS value (as a single value) before the participant came off treatment.
Time Frame: Baseline and the last KRAS value before the participant came off treatment, approximately 1- 8.2 months.
Measure: Mean (Standard Deviation); unit: copies
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
copies
  Baseline | 2584 (2242) | 1556 (480)
  Last recorded value | 6607 (6067) | 1542 (586)

10. Secondary Outcome: Overall Percentage Change (%) of Copies KRAS Wild Type Allele
Description: Overall ctDNA copy number measurements of KRAS wild type alleles in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant at baseline and last recorded value while on-treatment.
Time Frame: Approximately 1- 8.2 months.
Measure: Number; unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Percentage change | 156 | -1

11. Secondary Outcome: Mean Copy Number KRAS Mutant Type Allele in Circulating Tumor DNA (ctDNA)
Description: Mean ctDNA copy number measurements of KRAS mutant alleles in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples was determined at baseline and the last recorded value while on treatment.
Time Frame: Baseline and last recorded value while on treatment, approximately 1- 8.2 months.
Measure: Mean (Standard Deviation); unit: copies
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
copies
  Baseline | 3.33 (3.79) | 0 (0)
  On Treatment | 10.33 (15) | 1.6 (0.8)

12. Secondary Outcome: Overall Percentage Change of Copies KRAS Mutant Type Allele
Description: Overall ctDNA copy number measurements of KRAS mutant alleles in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant at baseline and last recorded value while on-treatment.
Time Frame: Approximately 1- 8.2 months.
Measure: Number; unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Percentage change | 210 | NA — The percentage was not calculable because the denominator had a value of 0.

13. Secondary Outcome: Percentage of KRAS Allele in Circulating Tumor DNA (ctDNA) That is Identified as Variant From Cell-free (cf) DNA
Description: This outcome measure is reporting the overall percentage of KRAS allele in circulating tumor DNA (ctDNA) that is identified as variant from cell-free (cf) DNA isolated from plasma samples between baseline and on-treatment.
Time Frame: Between baseline and last recorded value while on-treatment, approximately 1- 8.2 months.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Percentage
  Baseline | 7.5 (8.7891979156235) | 0 (0)
  Last recorded value | 9.33 (14.185281887302) | 8.5 (8.5)

14. Secondary Outcome: Overall Any Percent Change in (VAF, %), of KRAS Allele in Circulating Tumor Deoxyribonucleic Acid (ctDNA)
Description: Overall change in Variant Allele Fraction (VAF, %) of KRAS allele in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant between baseline and last recorded value while on-treatment
Time Frame: Approximately 1- 8.2 months.
Measure: Number; unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 6 | 2
Percentage change | 19.6 | 8.5

15. Secondary Outcome: Mean Change in Variant Allele Fraction (VAF, %) of KRAS in Participants Who Had No Measurable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) at Baseline
Description: Any change in Variant Allele Fraction (VAF, %) of KRAS allele in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant between baseline and while on-treatment in patients with no Mutant Fractional KRAS Abundency at baseline (VAF %, KRAS allele at baseline = 0% ).
Time Frame: Baseline and last recorded value while on-treatment, approximately 1- 8.2 months.
Population: Three out of 6 participants in dose level one and two out of 2 participants in dose level 2 had No Measurable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) at baseline.
Measure: Mean (Standard Deviation); unit: Variant Allele Fraction (VAF, %) of KRAS
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 3 | 2
Variant Allele Fraction (VAF, %) of KRAS
  Baseline | 0 (0) | 0 (0)
  Last recorded value | 0 (0) | 8.5 (8.5)

16. Secondary Outcome: Overall Percent Change in Variant Allele Fraction (VAF, %) of KRAS in Participants Who Had No Measurable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) at Baseline
Description: Overall change in Variant Allele Fraction (VAF, %) of KRAS allele in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant between baseline and while on-treatment in patients with no Mutant Fractional KRAS Abundency at baseline (VAF %, KRAS allele at baseline = 0% ).
Time Frame: Approximately 1- 8.2 months.
Population: as for outcome 15
Measure: Number; unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 3 | 2
Percentage change | 0 | 8.5

17. Secondary Outcome: Percentage Change of KRAS Allele in Circulating Tumor Deoxyribonucleic Acid (ctDNA) That is Identified as Variant From Cell-free (cf) DNA at Baseline and After Treatment
Description: This outcome measure is reporting the percentage of KRAS allele in circulating tumor DNA (ctDNA) that is identified as variant from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant between baseline and last recorded value after treatment in patients with detectable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) (Mutant Fractional KRAS Abundency at baseline and after treatment (VAF %), KRAS allele at baseline > 0%).
Time Frame: Baseline and last recorded value after treatment, approximately 1- 8.2 months.
Population: Two out of 6 participants in dose level one and 0 out of 2 participants in dose level 2 had detectable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) at baseline and after treatment
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 2 | 0
Percentage change
  Baseline | 18 (6) |
  Last recorded value | 28 (9) |

18. Secondary Outcome: Overall Percent Change in Variant Allele Fraction (VAF, %) of KRAS in Participants With Detectable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) at Baseline and After Treatment
Description: Overall change in Variant Allele Fraction (VAF, %) of KRAS allele in circulating tumor DNA (ctDNA) from cell-free (cf) DNA isolated from plasma samples determined from a single percentage change for the group rather than a percentage change for each participant with detectable KRAS Mutant Circulating Tumor Deoxyribonucleic Acid (ctDNA) between baseline and last recorded value after treatment.
Time Frame: Approximately 1- 8.2 months.
Population: as for outcome 17
Measure: Number; unit: Percentage change
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
Number analyzed (Participants) | 2 | 0
Percentage change | 60.9 |

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 25 months and 6 days.
Arm/Group | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/2
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily (N=6) | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily (N=2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: 75mg Selumetinib Sulfate Twice Daily (N=6) | 75mg Selumetinib Sulfate Twice Daily Follow/by 50mg TwiceDaily (N=2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 2 (10)
Alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 2 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 2 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 5 (6) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (General disorders) | 2 (2) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 4 (10) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (3) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03040986/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03040986/ICF_001.pdf